CLINICAL TRIAL: NCT03762629
Title: Effects of Exercise Training and Diet Restriction on Cardiovascular Function and Their Related Factors in Obese Chinese Children and Adolescents: an Intervention Study
Brief Title: Exercise and Diet Restriction on Cardiovascular Function in Obese Children and Adolescents
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Guangzhou Sport University (Other)
Responsible Party: Principal Investigator, Min Hu, Director of Guangdong Provincial Key Laboratory of Sports and Health Promotion, Guangzhou Sport University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Trial2017.1
Record Dates: First submitted 2017-07-02; First posted 2018-12-04 (Actual); Last update posted 2018-12-04 (Actual); Status verified 2018-12

CONDITIONS: Childhood Obesity; Adolescent Obesity
MeSH Terms: conditions — Pediatric Obesity | interventions — Exercise

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Obese intervention group (Experimental): Obese children were received exercise and diet intervention for 6 weeks.
  Interventions: Behavioral: Exercise
- Normal weight control group (No Intervention): Normal weight children were recruited as a control group without any intervention.

INTERVENTIONS:
Behavioral: Exercise — Subjects were provided with energy-restricted diets of 1300-2200 kcal/day based on weight. The energy percentages provided by protein, fat and carbohydrate were 20%, 20% and 60%, respectively, while energy distributions at breakfast, lunch and dinner were 30%, 40% and 30%, respectively. Subjects performed a series of endurance exercise such as bicycling, walking, running, dancing and ball games for 5 hour/day, supplemented with resistance exercise. Training interventions were performed 5-6 day/week for 6 weeks. The exercise program was designed to result in an energy expenditure of 1500-2500 kcal/day.
  Other Names: diet restriction
  Arms: Obese intervention group

SUMMARY:
Prevalence rates of childhood obesity have reached alarming levels. As childhood obesity may already be associated with serious comorbidities, obese adolescents are at significantly higher risk for obesity and increased morbidity and mortality during adulthood. Combined lifestyle interventions, which include regular physical activity and dietary restriction, have been shown to result in most significant improvements in cardiovascular function and their associated factors in the pediatric and adolescent population with obesity. The aim of this study is to investigate the effects of a combined exercise and diet intervention on cardiovascular function and their associated factors in obese children.

DETAILED DESCRIPTION:
Sixty obese children and adolescents will complete a 6-week program of exercise and diet intervention. Thirty normal-weight children and adolescents will be recruited as control group. Clinical characteristics, body composition, blood biochemistry, and circulating irisin levels of the subjects will be measured before and after 6-week intervention. Endothelial function will be assessed by a flow-mediated dilation test. Circulating exosome-derived miRNAs, exercise-induced epigenetic modifications, circulating irisin levels irisin concentration in plasma and arterial stiffness as well as cardiac autonomic function will be investigated before and after the 6-week intervention. Fecal samples were collected before and after the 6-week intervention for analysis of the compositional and functional changes in the human gut microbiota.

ELIGIBILITY:
Inclusion Criteria:

1. Participants aged 7-17 years
2. Participants satisfied the obesity diagnosis criteria is based on "Body mass index reference standards for the screening of overweight and obesity in Chinese children and adolescents" released in 2004, with cut-off points of p(95) for obesity

Exclusion Criteria:

1. Metabolic disease
2. Gastrointestinal disease
3. Cardiac disease
4. Taking medications which affected energy expenditure
5. Losing weight in the past three months whether by diet, taking weight-loss medication or more physical exercise than normal

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 90 (Estimated)
Dates: Start 2017-07-01 (Actual); Primary Completion 2018-12-31 (Estimated); Study Completion 2018-12-31 (Estimated)

PRIMARY OUTCOMES:
Change from flow-mediated dilation (FMD) at 6 weeks | before and after the 6-week intervention
  for brachial endothelial function assessment

SECONDARY OUTCOMES:
Change from circulating exosome-derived miRNAs at 6 weeks | before and after the 6-week intervention
  exosome-secreted miRNA levels in plasma
Change from circulating irisin levels at 6 weeks | before and after the 6-week intervention
  irisin concentration in plasma
Change from pulse wave velocity at 6 weeks | before and after the 6-week intervention
  for arterial stiffness assessment
Change from heart rate variability at 6 weeks | before and after the 6-week intervention
  for cardiac autonomic function assessment

OTHER OUTCOMES:
Change from the composition of gut microbiota at 6 weeks | before and after the 6-week intervention
  the composition of gut microbiota in fecal samples
Change from short chain fatty acids (SCFAs) concentractions at 6 weeks | before and after the 6-week intervention
  short chain fatty acids (SCFAs) concentractions in fecal samples

CONTACTS AND LOCATIONS:
Overall Officials: Min Hu, PhD, Principal Investigator — Guangzhou Sport University
Locations (1):
- Guangzhou Sport University, Guangzhou, Guangdong, China

REFERENCES:
- [Derived] Huang J, Liao J, Fang Y, Deng H, Yin H, Shen B, Hu M. Six-Week Exercise Training With Dietary Restriction Improves Central Hemodynamics Associated With Altered Gut Microbiota in Adolescents With Obesity. Front Endocrinol (Lausanne). 2020 Dec 7;11:569085. doi: 10.3389/fendo.2020.569085. eCollection 2020. PMID 33365012
- [Derived] Liao J, Huang J, Wang S, Xiang M, Wang D, Deng H, Yin H, Xu F, Hu M. Effects of exercise and diet intervention on appetite-regulating hormones associated with miRNAs in obese children. Eat Weight Disord. 2021 Mar;26(2):457-465. doi: 10.1007/s40519-020-00869-9. Epub 2020 Feb 18. PMID 32072570